CLINICAL TRIAL: NCT01947179
Title: Development and Evaluation of a Brief, Suicide Prevention Intervention Reducing Anxiety Sensitivity
Brief Title: Cognitive Anxiety Sensitivity Treatment for Suicide
Acronym: CAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Norman Schmidt, Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 03969
Record Dates: First submitted 2013-09-12; First posted 2013-09-20 (Estimated); Last update posted 2013-09-26 (Estimated); Status verified 2013-09

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical Health Training (No Intervention): The Physical Health Training condition will include information on the importance and benefits of a healthy lifestyle. Additionally, the program will discuss guidelines for a healthy lifestyle including information on diet, water consumption, exercise, and sleep.
- Anxiety Risk Reduction (Experimental): The anxiety risk reduction intervention will include psychoeducation focused on the nature of stress and its effect on the body. Interoceptive exposure exercises that were designed to correct the conditioned fear of bodily sensations will be explained and practiced.
  Interventions: Behavioral: Anxiety Risk Reduction

INTERVENTIONS:
Behavioral: Anxiety Risk Reduction — Involves psychoeducation and interoceptive exposure exercises
  Arms: Anxiety Risk Reduction

SUMMARY:
The purpose of this study is to test the effectiveness and usability of a computer-based treatment for mood and anxiety relevant risk factors. The target of the treatment is related to cognitive stress, which has been shown to be associated with several negative mental health outcomes such as suicidal ideation, substance use disorders, and Post-Traumatic Stress Disorder.

DETAILED DESCRIPTION:
CAST is a newly developed computerized treatment targeting specific risk factors associated with PTSD, substance use, anxiety, and suicide. Eligible individuals will be randomized to one of two conditions. In both conditions, participants will complete various self-report questionnaires and a computerized presentation. Additionally, all participants will be asked to complete a one month follow-up appointment.

ELIGIBILITY:
Inclusion Criteria:

* At or above the community sample mean on the ASI
* English speakers
* 18 years of age or older

Exclusion Criteria:

* Significant medical illness
* Current substance dependence
* Current or past psychotic-spectrum disorders
* Uncontrolled bipolar disorder
* Serious suicidal intent that warranted immediate medical treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2011-09; Primary Completion 2013-01 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Anxiety Sensitivity Index (ASI) | Month one follow-up
  The ASI is a 16-item self-report measure of anxiety sensitivity. Each item consists of a possible negative consequence of anxiety symptoms. The scale assesses three AS subfactors including cognitive, physical, and social concerns. The measure has shown good psychometric properties.

SECONDARY OUTCOMES:
Beck Suicide Scale (BSS) | Month one follow-up
  The BSS is a 21-item widely used self-report measure assessing a broad spectrum of behaviors and attitudes related to suicide risk, including suicidal ideation and past suicide attempts. It has demonstrated strong reliability and validity.

OTHER OUTCOMES:
Posttraumatic Diagnostic Scale (PDS) | Month one follow-up
  The PDS is a self-report measure used to assess the severity of posttraumatic stress symptoms during the past month. The measure was designed based on Diagnostic and Statistical Manual-IV criteria. Respondents report if they have experienced any of 12 traumatic events, including an "other" category, and then indicate which event was the most disturbing. Additionally, respondents rate the frequency of 17 PTSD symptoms experienced in the past month in relation to the most disturbing event they endorsed. The PDS has excellent psychometric properties and can be used as a continuous measure of PTSD symptom severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Florida State University, Tallahassee, Florida, United States